CLINICAL TRIAL: NCT00763828
Title: Can Hypothermia be Incorporated Into Primary Angioplasty for Heart Attack?
Acronym: CHIPAHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Life Recovery Systems (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRS-01-07-01
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: Myocardial Infarction; Hypothermia, Induced
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Hypothermia | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ThermoSuit-Induced Patient Cooling (Experimental): The Life Recovery Systems ThermoSuit System will be used to cool STEMI patients under conditions of conscious sedation.
  Interventions: Device: Life Recovery Systems ThermoSuit

INTERVENTIONS:
Device: Life Recovery Systems ThermoSuit — Hypothermia induction (cooling to 32 to 34 degrees C core temperature) using the Life Recovery Systems ThermoSuit System (a device which cools patients using direct skin contact with cold water) followed by PCI (percutaneous coronary intervention) and maintenance of hypothermia for 3 hours following PCI.
  Other Names: Life Recovery Systems ThermoSuit(R) System

SUMMARY:
The hypothesis of this study is that consciously sedated patients suffering from ST-elevation myocardial infarction can be rapidly and safely cooled to a state of therapeutic hypothermia (32 to 34 degrees C) using the LRS ThermoSuit System prior to percutaneous coronary intervention.

DETAILED DESCRIPTION:
This clinical study will investigate the safety and feasibility of cooling heart attack (STEMI) patients with the LRS (Life Recovery Systems)ThermoSuit System, a cooling device which uses the principle of cold water immersion to rapidly reduce patient temperature. The study will enroll a total of up to 20 patients, and will be a cooperative effort between LRS and LSU Health Sciences Center - Shreveport.

The study is being conducted under an IDE (Investigational Device Exemption) that was granted to LRS by FDA (G070141). The primary goal of this trial is to demonstrate the feasibility of cooling AMI patients pre-reperfusion with the ThermoSuit cooling device. The safety of this treatment will be determined by review of a composite of serious adverse events.

Consciously sedated patients will be cooled after entry into the emergency room and prior to percutaneous coronary intervention in the catheterization laboratory. It is hypothesized that the ThermoSuit System will enable cooling of the patient to 34ºC after a treatment of 30 minutes or less. Previous research has suggested that cooling of ST-elevation myocardial infarction patients before coronary reperfusion could result in a significant reduction in myocardial infarct size.

If successful, this study will lead to a pivotal clinical study to investigate the potential for the ThermoSuit cooling treatment to reduce myocardial infarct size. The ultimate goal of these studies is to determine the safety and effectiveness of the use of the ThermoSuit device for the treatment of AMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Duration of MI symptoms ≥ 30 minutes to ≤ 6 hours.
* ST-segment elevation of ≥ 1mm or more in two or more contiguous leads.
* Eligible for PCI.
* Willingness of patient or legal guardian to provide written, informed consent.
* Patient dimension criteria:
* Height: 147-190 cm (58 - 75 in)
* Width: ≤73 cm (29 in) (elbow to elbow)

Exclusion Criteria:

* Cardiac arrest or previous MI within one month.
* Administration of thrombolytics.
* Cardiogenic shock (systolic blood pressure (SBP) < 80 mmHg for > 30 minutes or SBP < 100 mmHg on vasopressors or IABP) in the absence of bradycardia or other correctable causes.
* Known hypersensitivity to hypothermia including Raynaud's disease or cryoglobulinemia.
* Severe allergy or contraindication to aspirin, Plavix, heparin, or contrast media which cannot be adequately pre-medicated.
* History of bleeding diathesis or coagulopathy or refusal of blood transfusions.
* Pregnancy.
* Known hypersensitivity midazolam, meperidine, buspirone, or magnesium sulfate.
* Current enrollment in another clinical trial (other than registry).
* Temperature < 35°C on admission to Emergency Department.
* Recent (< 1 week) surgical incisions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-28 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of use of cooling device as determined by ability and time to achieve target temperature and ease of maintaining temperature in therapeutic range (32 to 34°C) for three hours following removal of patient from ThermoSuit. | Four hours
Primary safety endpoint: composite of serious adverse events including: death, re-infarction, ischemia-driven TVR, pneumonia, sepsis, arrhythmia, bleeding, stroke, and renal failure. | 30 days post-hospital discharge

SECONDARY OUTCOMES:
Major adverse cardiac events at 30 days as defined by death or non-fatal re-infarction. c. Ischemia-driven target vessel revascularization. | 30 days post-hospital discharge
Myocardial infarct size at 30 days as measured by 99mTc-sestamibi SPECT imaging. | 30 days post-hospital discharge
Safety, including all-cause mortality, cardiac, vascular, and hematological complications. | 30 days post-hospital discharge
Adverse events associated with conscious sedation. | 30 days post-hospital discharge
Arterial blood pressure and heart rate every 5 minutes from the baseline just before the start of cooling until 30 minutes after cooling has started. | One hour
Door to balloon time. | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Freedman, M.D., Study Chair — Life Recovery Systems
Locations (1):
- UTHSCSA, San Antonio, Texas, United States